CLINICAL TRIAL: NCT05650502
Title: Impact of Seasonal Malaria Chemoprevention on the Acquisition and Maintenance of Immunity Against Malaria Among Children in Northern Benin
Brief Title: Impact of Seasonal Malaria Chemoprevention on Immunity Against Malaria Among Children in Northern Benin
Acronym: ISAMIMA
Status: Completed | Type: Observational
Sponsor: Université de Parakou (Other)
Collaborators: Institut de Recherche pour le Developpement (Other Government); University of Copenhagen (Other); University of Ghana (Other); Institut de Recherche Clinique du Bénin (IRCB) (Unknown); Hôpital Cochin (Other)
Responsible Party: Principal Investigator, Azizath Moussiliou, Assistant Professor, Université de Parakou
Other Study IDs: University of Parakou
Record Dates: First submitted 2022-12-04; First posted 2022-12-14 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Plasmodium Malariae Infection; SMC; Immune System Disease
Keywords: Seasonal malaria chemoprevention; Malaria; Children; Anti PfEMP1
MeSH Terms: conditions — Immune System Diseases; Malaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ISC (ISAMIMA children group-Cobly): This group included children from 6 to 59 months living in Cobly and receiving the SMC treatment. The treatment is administered for three consecutives days for 4 months (from july to october).
  For children under 12 months: one dose of SP 250/12.5mg on day 1 AQ 75mg once daily for 3 days For children from 12 to 59 months: one dose of SP 500/25mg on day 1 AQ 150 mg once daily for 3 days A monthly visit was planned for monitoring during the follow up. Sample was collected in jun, september, january and April.
  Interventions: Drug: saisonal malaria chimoprevention
- IST (ISAMIMA children group-Tchaourou): This group included children from 6 to 59 months living inTchaourou and who did not receiving the SMC treatment.
  A monthly visit was planned for monitoring during the follow up. Sample was collected in jun, september, january and April.
  Interventions: Drug: saisonal malaria chimoprevention

INTERVENTIONS:
Drug: saisonal malaria chimoprevention — Investigate the impact of saisonal malaria chimoprevention on children anti PfEMP1 construction and maintenance and their succeptibility to malaria infection

SUMMARY:
This study aims to evaluate the effects of SMC (Seasonal malaria chemoprevention) with Sulfadoxine-Pyrimethamine (SP) and Amodiaquine (AQ) on the evolution of anti-malarial immunity of children and their susceptibility to malarial infection.

This is a cross-sectional study on children aged 6 to 59 months with/without SMC in two villages in northern Benin. Sociodemographic and clinical data as well as repeated blood samples will be collected from 440 children (before, during and after treatment). Samples will be analyzed using a Luminex assay to investigate antibody responses to MSP (merozoite surface protein) , Glurp (Glutamate-Rich Protein) and a panel of PfEMP1. qPCR (quantitative polymerase chain reaction) will be used to detect the prevalence of malaria at this period and parasites infecting children will be characterize during the follow up.

DETAILED DESCRIPTION:
Study location and population The study was conducted in parallel in two different sites, the health districts of Cobly and Tchaourou (two villages) located in northern Benin. These two districts have been chosen based on the Ministry of Health's programming for the implementation of SMC. The two sites were very similar in terms of malaria transmission characteristics and epidemiology, with the difference that SMC was implemented in Cobly but not in Tchaourou. Participants will be informed on the importance of SMC. A written informed consent was collected from parent or guardian of each child. Participation was entirely voluntary.

Study Design and procedures This is a case control study focuses on the follow-up over 12 months of children aged 6 to 59 months in northern Benin. The study was conducted in collaboration with National Malaria Control Program (NMCP). Demographic data generated by the NMCP had allow us for a random selection of children from random households. In both intervention and control sites, equal numbers of children were included. The study team visited each selected household to inform members. A monthly visit has been set up for monitoring. Children of consenting parents or guardians were recruited and parents/guardians were taken through a questionnaire administered by the researcher or an assistant (clinician). 1 ml of peripheral venous blood was collected into collection tubes and transferred to the Center for Expertise and Enhancing Research in Epidemiology and Public Health (CEEREPH) at the University of Parakou where a blood smear was prepared from each sample. Fifty microliters of blood have been transferred to Whatman 3MM filter paper and stored at room temperature for DNA extraction. The remaining whole blood have been centrifuged. The plasma and red blood cells were aliquoted. Samples was collected at 4 times during the 12 months follow-up period. The first samples were collected at the beginning of SMC implimentation (before children receive the first SMC dose), the second blood sample were collected at the day of the third dose of SMC, the third, at three month after the last dose of SMC and the fourth, six months after the last dose of SMC).

Malaria prevalence Thick and thin blood smears whave been prepared from all samples at all four times. Thick smears will be fixed in methanol. All slides were air dried and stained using Giemsa stain 3% for 45-60 min. Once dry, the stained thick and thin blood films were examined microscopically using a routine procedure. Parasite densities was recorded as the number of parasites/μl of blood assuming an average leukocyte count of 8,000/μl of blood. Dried blood spots were air dried and stored individually in small Ziploc bags with a desiccant. Plasmodium spp detection was performed using a real time polymerase chain reaction (qPCR).

Anti-PfEMP1 antibody response Plasmodium falciparum-encoded variant surface antigens (VSA) are expressed on the surface of infected erythrocytes (IE) and mediate binding to a range of endothelial cell receptors. The best characterized VSA are the var gene-encoded P. falciparum erythrocyte membrane protein 1 (PfEMP1) family in two exon units. Exon I codes for the extracellular and variable part of the protein as well as a transmembrane region and Exon II encodes the intracellular and relatively conserved acidic terminal segment (ATS). The most variable part of the protein contains a N-terminal segment followed by segments composed of three domain types; Duffy binding-like domains (DBL-domains): Cysteine-rich inter-domain regions (CIDRs) and C2. In this study, a panel of plasma antibody was quantified using microsphere bead-coupled proteins comprising 28 P. falciparum-derived antigens and tetanus toxoid, using the Luminex platform. The panel includes VAR2CSA (the VSA associated to placental malaria) and 25 HIS-tagged CIDR proteins representing all three main groups of PfEMP1, merozoite surface protein 1 (MSP1) and apical membrane antigen 1 (AMA1).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 59 months
* Have been selected and accepted to receive SMC treatment (SP-AQ) in the intervention site and not in the control site
* Be able to take drugs

Exclusion Criteria:

* Child whose parents will no longer consent at some point in the study for one reason or another
* Children suffering from a chronic disease
* Intolerance to certain drugs

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who meet the inclusion and exclusion criteria, living in the communes of Cobly and Tchaourou located in northern Benin, whether or not they have received Saisonal malaria chimotreatment, will be recruited.
Sampling Method: Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Efficiency of Seasonal malaria chemoprevention | January 2023
  Malaria prevalence during the intervention

SECONDARY OUTCOMES:
Impact of Seasonal malaria chemoprevention | June 2023
  Hospital frequency rate of children

CONTACTS AND LOCATIONS:
Overall Officials: Nicaise TIUKUE NDAM, Professor, Study Chair — Institut régional de développement IRD (UMR261); Adrian LUTY, Professor, Study Chair — Institut régional de développement IRD (UMR261)
Locations (1):
- Azizath MOUSSILIOU, Parakou, Benin

IPD SHARING:
Plan to Share IPD: No
Protocol and the informed consent will be shared with other researchers